CLINICAL TRIAL: NCT00535171
Title: Venous Thromboembolism Taskforce Audit Program
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Other Study IDs: DIREG_L_01927
Record Dates: First submitted 2007-09-25; First posted 2007-09-26 (Estimated); Last update posted 2010-01-22 (Estimated); Status verified 2010-01

CONDITIONS: Venous Thrombosis
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
To determine the effect of an interventional campaign run by a dedicated "VTE Nurse Educator" over a 6-month period and the effect on prophylaxis rates.

To determine the proportion of medically admitted patients with risk factors for VTE.

To assess and compare the use of venous thromboembolism (VTE) prophylaxis in hospitalized medical patients versus recommendations and current guidelines.

To determine the patient characteristics of those deemed to be at risk of VTE. To determine the proportion of patients receiving appropriate thromboprophylaxis for their risk.

To determine the type and duration (where possible) of prophylaxis used.

ELIGIBILITY:
Inclusion Criteria:

* Hospital admission for an acute illness with an in-patient hospital stay of 3 days or more.

Exclusion Criteria:

* Patients who have undergone any type of surgery during current admission
* Patients who are admitted to a ward or department that is excluded from this study e.g psychiatric, paediatric, maternity, intensive care unit, coronary care unit.
* Prior enrollment in this protocol during current admission
* Prior enrollment in a VTE study involving pharmaceutical or mechanical treatment within last 90 days.
* Admission for suspected or diagnosed deep vein thrombosis

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Venous thromboembolism in medical patients bedridden due to acute illness.
Sampling Method: Probability Sample
Enrollment: 8764 (Actual)
Dates: Start 2007-06; Primary Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Howard, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Macquarie Park, Australia